CLINICAL TRIAL: NCT05048797
Title: An Open-label, Randomized, Multicenter, Phase 3 Study to Assess the Efficacy and Safety of Trastuzumab Deruxtecan as First-line Treatment of Unresectable, Locally Advanced, or Metastatic NSCLC Harboring HER2 Exon 19 or 20 Mutations (DESTINY-Lung04)
Brief Title: A Study to Investigate the Efficacy and Safety of Trastuzumab Deruxtecan as the First Treatment Option for Unresectable, Locally Advanced/Metastatic Non-Small Cell Lung Cancer With HER2 Mutations
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D967SC00001; 2023-503674-20-00 (Registry Identifier: CTIS); 2021-000634-33 (EudraCT Number)
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Keywords: DS-8201a; HER2 exon 19 or 20 mutations; ERBB2 gene (coding for the HER2 protein); T-DXd; Trastuzumab Deruxtecan; Locally advanced and unresectable non-squamous NSCLC; Metastatic non-squamous NSCLC; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trastuzumab deruxtecan; Cisplatin; Carboplatin; pembrolizumab; Pemetrexed

STUDY DESIGN:
Intervention Model Description: This study consists of two open-label treatment arms:
  Arm 1: Trastuzumab Deruxtecan Arm 2: Standard of Care treatment (platinum, pemetrexed and pembrolizumab)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Trastuzumab Deruxtecan (T-DXd)
  Interventions: Drug: Trastuzumab Deruxtecan
- Arm 2 (Active Comparator): Standard of Care Treatment (platinum, pemetrexed and pembrolizumab)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pembrolizumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Trastuzumab Deruxtecan administered by intravenous infusion
  Other Names: DS-8201a; T-DXd
  Arms: Arm 1
Drug: Cisplatin — Investigator's choice of platinum chemotherapy (cisplatin) administered by intravenous infusion
  Arms: Arm 2
Drug: Carboplatin — Investigator's choice of platinum chemotherapy (carboplatin) administered by intravenous infusion
  Arms: Arm 2
Drug: Pembrolizumab — Pembrolizumab administered by intravenous infusion
  Arms: Arm 2
Drug: Pemetrexed — Pemetrexed administered by intravenous infusion
  Arms: Arm 2

SUMMARY:
DESTINY-Lung04 will investigate the efficacy and safety of Trastuzumab Deruxtecan (T-DXd) versus Standard of Care (SoC) as first-line treatment of Non-Small Cell Lung Cancer (NSCLC) with HER2 Exon 19 or 20 mutations

DETAILED DESCRIPTION:
Eligible participants will be those diagnosed with unresectable, locally advanced or metastatic histologically documented non-squamous NSCLC with HER2 exons 19 or 20 mutations and who are treatment-naïve for palliative intent systemic therapy for locally advanced or metastatic disease.

The study aims to evaluate the efficacy, safety and tolerability of trastuzumab deruxtecan as first-line treatment of Non-Small Cell Lung Cancer (NSCLC) as compared with Standard of Care treatment (Investigator's choice of cisplatin or carboplatin + pembrolizumab + pemetrexed). This study aims to see if trastuzumab deruxtecan allows patients to live longer without the cancer getting worse or simply to live longer, compared to patients receiving standard of care treatment. This study is also looking to see how the treatment and the cancer affects patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 18 years of age
* Locally advanced and unresectable NSCLC, not amenable to curative therapy, or metastatic disease
* Histologically documented non-squamous NSCLC with HER2 mutation in exons 19 or 20 by tissue NGS or ctDNA
* Treatment-naïve for palliative intent systemic therapy for locally advanced or metastatic disease
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Measurable disease assessed by Investigator based on RECIST 1.1
* Protocol-defined adequate organ function including cardiac, renal, hepatic function
* ECOG 0-1
* Having tumour tissue available for central testing

Exclusion Criteria:

* Tumors with targetable alterations to EGFR (or other targetable mutations including but not limited to ALK, if routinely tested as a targetable alteration with approved available therapy)
* Any untreated brain metastases, including asymptomatic or clinically inactive brain metastases
* Active autoimmune or inflammatory disorders
* Medical history of myocardial infarction within 6 months prior to randomization
* History of non-infectious pneumonitis/ILD, current or suspected ILD
* Lung-specific intercurrent clinical significant severe illness
* Contraindication to platinum-based doublet chemotherapy or pembrolizumab

Ages: 18 Years to 123 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) | Until progression or death, assessed up to approximately 12 months
  Defined as time from randomization until progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR), or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Until death, assessed up to approximately 28 months.
  Defined as time from randomization until the date of death due to any cause.
Progression Free Survival (PFS) by investigator assessment | Until progression, assessed up to approximately 12 months
  Defined as time from randomization until progression per RECIST 1.1 as assessed by the investigator, or death due to any cause.
Objective Response Rate (ORR) | Until progression, assessed up to approximately 12 months
  Defined as the proportion of participants who have a complete response (CR) or partial response (PR) as assessed by Blinded Independent Central Review (BICR) and investigator according to RECIST 1.1
Duration of Response (DoR) | Until progression, assessed up to approximately 12 months
  Defined as the time from the date of first documented response until date of documented progression as assessed by Blinded Independent Central Review (BICR) and investigator assessment according to RECIST 1.1.
Time to second progression or death (PFS2) | Assessed up to approximately 20 months
  Defined as the time from randomization until second progression on next-line of treatment as assessed by investigator at the local site using assessments conducted per local standard clinical practice, or death due to any cause.
Landmark analysis of PFS (PFS12) | Assessed up to approximately 12 months
  Defined as proportion of participants alive and progression-free at 12 months, as assessed by Blinded Independent Central Review (BICR) and investigator.
Landmark analysis of OS (OS24) | Assessed up to approximately 24 months
  Defined as proportion of participants alive at 24 months
Central Nervous System (CNS) - Progression Free Survival (PFS) | Until CNS progression or death, assessed up to approximately 12 months
  Defined as time from randomization until Central Nervous System (CNS) progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR) or death due to any cause in the absence of CNS progression.
Safety and tolerability of T-DXd versus Standard of Care treatment | Until progression or death, assessed up to approximately 28 months
  Assessed by the occurrence of AEs, SAEs, and changes from baseline in laboratory parameters, vital signs, ECG, and ECHO/MUGA scan results.
Pharmacokinetics (PK) of T-DXd, total anti-HER2 antibody and DXd in serum | Up to cycle 4, approximately 12 weeks
  Serum concentration of T-DXd, total anti-HER2 antibody and DXd.
Immunogenicity of T-DXd | Until progression, assessed up to approximately 13 months
  Presence of anti-drug antibodies (ADAs) for T-DXd.
Patient-reported pulmonary symptoms associated with Non-Small Cell Lung Cancer | Until progression, assessed up to approximately 13 months
  Time to sustained deterioration in pulmonary symptoms (cough, dyspnea, chest pain) while on treatment using the Non-Small Cell Lung Cancer-Symptom Assessment Questionnaire (NSCLC-SAQ).
Patient-reported tolerability of T-DXd described using symptomatic AEs | Until progression, assessed up to approximately 13 months
  Symptomatic AEs: Descriptive summary of the proportion of participants reporting symptomatic AEs while on treatment, as assessed by the Patient-reported outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) and items from the European Organisation for Research and Treatment of Cancer (EORTC) Item Library.
Patient-reported tolerability of T-DXd described using overall side-effect bother | Until progression, assessed up to approximately 13 months
  Overall side-effect bother: Descriptive summary of the proportion of participants reporting overall side-effect bother on the Patient's Global Impression of Treatment Tolerability (PGI-TT) while on treatment.
Patient-reported tolerability of T-DXd described using physical function | Until progression, assessed up to approximately 13 months
  Physical Function: The proportion of participants with maintained or improved physical function while on treatment, based on the European Organisation for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC-QLQ-C30) physical functioning scale.

CONTACTS AND LOCATIONS:
Locations (119):
- United States (19):
  - Research Site, Anchorage, Alaska
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Basking Ridge, New Jersey
  - Research Site, Middletown, New Jersey
  - Research Site, Montvale, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Commack, New York
  - Research Site, Harrison, New York
  - Research Site, New York, New York
  - Research Site, Uniondale, New York
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
- Austria (2):
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Ghent
  - Research Site, Leuven
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Natal
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Uberlândia
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, Brampton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (20):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yangzhou
- Research Site, Vejle, Denmark
- France (8):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Oldenburg
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Jordan
- India (5):
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, Nashik
- Italy (6):
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Roma
  - Research Site, Verona
- Japan (13):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kashiwa
  - Research Site, Matsuyama
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Yokohama
  - Research Site, Yonago-shi
- Research Site, Mexico City, Mexico
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Nijmegen
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Olsztyn
  - Research Site, Przemyśl
  - Research Site, Warsaw
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (4):
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Research Site, Çankaya
  - Research Site, Edirne
  - Research Site, Izmir
  - Research Site, Kadıkoy/Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/304247